CLINICAL TRIAL: NCT04382339
Title: Effectiveness of Sofosbuvir/Pegylated-interferon Plus Ribavirin in Treatment of Hepatitis C Virus Genotype 4 Patients
Brief Title: Sofosbuvir/Pegylated-interferon Plus Ribavirin With HCV Genotype 4
Acronym: HCV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohammed Abdel-Gabbar, Ph.D, Associate Prof, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOF-PEG
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Hepatitis C Virus Infection
Keywords: HCV genotype 4; sofosbuvir; Peg-interferon α-2; ribavirin; Egyptian patients; Experinced; Naive
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment-naive (Active Comparator): Naive Egyptians having HCV GT4 received SOF, RBV, and PegINFα-2 once weekly for 12 weeks
  Intervention: 1 DDA: Sofosobuvir (SOF) plus Ribavirin (RBV) and pegylated-interferon (PegINFα-2)
  Interventions: Drug: SOF/RBV/PegINFα-2
- Treatment-experienced (Active Comparator): Experienced Egyptians having HCV GT4 received SOF, RBV, and PegINFα-2 once weekly for 12 weeks
  Intervention: 1 DDA: Sofosobuvir (SOF) plus Ribavirin (RBV) and pegylated-interferon (PegINFα-2)
  Interventions: Drug: SOF/RBV/PegINFα-2

INTERVENTIONS:
Drug: SOF/RBV/PegINFα-2 — SOF: block the hepatitis C NS5B protein. RBV: a nucleoside inhibitor PegINFα-2: chemically modified form of the standard interferon that treats hepatitis C

SUMMARY:
This study aims to assess the efficacy and safety of sofosbuvir (SOF) with pegylated interferon (PegINF)/ribavirin (RBV) for chronic HCV GT4 participants

DETAILED DESCRIPTION:
Between March 2015 and November 2015, 99 participants (59 naïve and 40 experienced) infected with HCV GT4 were enrolled in the study. Eligible participants received daily oral 400 mg SOF ( (Sovaldi, Gilead Sciences, Inc., USA), RBV (Copegus, Roche, Europe) based on body weight: < 75 kg, 1000 mg; ≥75 kg, 1200 mg), the dose modified according to participants tolerability, plus 180 μg PegINFα-2 once weekly for 12 weeks.

Experienced participants included participants with a prior relapse or a null response to PegINF/RBV therapy.

ELIGIBILITY:
Inclusion Criteria:

The study population consisted of treatment-naïve and treatment-experienced adults patients aged 20-65 with HCV RNA level > 10,000 IU/ml.

Experienced participants included those with a prior relapse or a null response to PegINF/RBV therapy.

-

Exclusion Criteria:Participants with one or more of

* HCV coinfected with hepatitis B virus (HBV)
* human immunodeficiency virus (HIV)
* had any liver disease other than chronic HCV GT4 infection.
* had a history of liver decompensation
* serum a-fetoprotein (AFP) > 100 ng/ml
* evidence of hepatocellular carcinoma
* major severe illness such as respiratory, renal, heart failure or autoimmune disease
* non-compliance with treatment.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12) in Each Treatment Arm SVR12 | 12 weeks after last dose
  SVR12 was defined as hepatitis C virus ribonucleic acid (HCV RNA) < 15 IU/m 12 weeks after the last dose of drugs.
Number of Participants With Adverse Events in Each Treatment Arm | Screening until 30 days after last dose
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or i clinical investigation after administering a pharmaceutical drugs serious adverse event (SAE) is an event that results in death, life-threatening, requires hospitalization, or significant disability/incapacity

SECONDARY OUTCOMES:
Percentage of Participants With Viral relapse | 12 weeks after last dose
  Viral relapse was HCV RNA undetectable at EOT, but detectable HCV RNA > 15 IU/ml levels 12 weeks after planned EOT.
Percentage of Participants With On-treatment Virologic Failure | up tp 24 weeks
  On-treatment virologic failure was defined as quantifiable HCV RNA throughout the entire treatment period with HCV RNA greater than 15 IU/ml

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Abdel-Gabbar, Ass. Prof, Principal Investigator — Biochemistry Dep., Faculty of Science, Beni-Suef University, P.O. Box 52621

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdel-Moneim A, Abood A, Abdel-Gabaar M, Zanaty MI, Ramadan M. Effectiveness of sofosbuvir/pegylated-interferon plus ribavirin in treatment of hepatitis C virus genotype 4 patients. Clin Exp Hepatol. 2018 Sep;4(3):191-196. doi: 10.5114/ceh.2018.78123. Epub 2018 Sep 10. PMID 30324144
- See also: The link clarify the effectiveness of sofosbuvir/pegylated-interferon plus ribavirin in treatment of hepatitis C virus genotype 4 patients — https://www.termedia.pl/Effectiveness-of-sofosbuvir-pegylated-interferon-plus-ribavirin-in-treatment-of-hepatitis-C-virus-genotype-4-patients,80,33652,0,1.html